CLINICAL TRIAL: NCT06011681
Title: The Proactive Screening and Diagnosis of Mild Cognitive Impairment and Depression in Patients Ages 60 and Over: An Implementation Study
Brief Title: The Rapid Diagnosis of MCI and Depression in Patients Ages 60 and Over
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Miro Health (Other)
Responsible Party: Sponsor
Other Study IDs: MH202206MCILLD
Record Dates: First submitted 2022-08-23; First posted 2023-08-25 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Depression; Mild Cognitive Impairment
MeSH Terms: conditions — Depression; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Depression: Seniors diagnosed with late life depression or with a concern of late life depression.
- Mild cognitive impairment: Seniors with self-reported decline in cognitive function or with a diagnosis of mild cognitive impairment.
- Healthy controls: Seniors with no neurological or psychiatric symptoms or conditions.

SUMMARY:
Mild cognitive impairment (MCI) leading to Alzheimer's disease and related disorders (ADRD) represents a significant health and economic burden of the rapidly expanding senior population. The accurate detection and diagnosis of MCI and its common comorbidity, late-life depression (LLD), is essential for prolonging patient quality of life and developing advancements in research and treatment options. The purpose of the proposed program is to refine Miro Health's A.I. to accurately detect, differentiate and diagnose MCI and LLD.

ELIGIBILITY:
Inclusion Criteria:

* LLD: Age 60 or over; diagnosis of LLD or symptoms consonant with LLD; PHQ-9 score from 15 to 27
* MCI: Age 60 or over; diagnosis of MCI or self-reported insidious onset and continued worsening of cognitive decline; intact activities of daily living
* HC: Age 60 or over

Exclusion Criteria:

* Age 59 or younger; history of unresolved neurological or psychiatric conditions; current medications known to affect cognition; history of substance abuse; unable to perform activities of daily living; change in employment status due to condition

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include healthy, worried well, depressed, and mild cognitively impaired seniors from multiple, disparate U.S. geographic regions.
Sampling Method: Non-Probability Sample
Enrollment: 960 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Measure usability of Miro Health assessments (iOS and Android) for patients | Year 1, Q3 - Year 2, Q2
  Measure the (a) time point 1 in-assessment drop-out rate; and (b) the rate of lost-to-time-point-2-followup at 12 months.
Measure acceptability of Miro Health assessments (iOS and Android) for patients | Year 1, Q3 - Year 2, Q2
  Measure the participant preference for pencil-paper test or Miro Health Mobile Assessment

SECONDARY OUTCOMES:
Measure domain score correlations of pencil-paper tests and Miro Health Mobile Assessment | Year 1, Q1 - Year 2, Q2
  Pairwise correlations greater than 0.8 and statistically significantly greater than 0.7 will be considered successful.

OTHER OUTCOMES:
Measure relevance of algorithms in separating depressed, MCI, and healthy control groups | Year 1, Q1 - Year 2, Q2
  Measure AUROC for: MCI vs healthy control; MCI vs aMCI; MCI vs depression; aMCI vs healthy control; aMCI vs depression; depression vs healthy control; and MCI + depression vs healthy control. AUROC equal to or greater than 0.84 is considered successful.

CONTACTS AND LOCATIONS:
Overall Officials: Shenly Glenn, BS, Principal Investigator — Miro Health
Locations (2):
- United States (2):
  - Miro Health, Sacramento, California
  - Miro Health, Miami, Florida